CLINICAL TRIAL: NCT07290153
Title: Prospective Observational Study of Psychological State, Immunotherapy Response, and Multi-Omics Features in Triple-Negative Breast Cancer
Brief Title: Psychological State, Immunotherapy Response, and Multi-Omics Signatures in TNBC
Acronym: SCHBCC-N0105
Status: Recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Professor, Fudan University
Other Study IDs: SCHBCC-N0105
Record Dates: First submitted 2025-12-06; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer Female NOS; General Anxiety Disorder; Depressive Disorder
Keywords: Breast Cancer
MeSH Terms: conditions — Generalized Anxiety Disorder; Depressive Disorder; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — This study will collect serial biospecimens and imaging data during neoadjuvant immunotherapy. Peripheral blood samples will be obtained for cytokine and immune profiling. Saliva samples will be collected for cortisol assessment. Surgical tumor specimens will be obtained at the time of definitive surgery. Radiological imaging at each treatment evaluation timepoint will also be collected. These materials will be used to analyze the association between psychological status, immune activation, and treatment efficacy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chemotherapy plus PD-1/PD-L1 inhibitor (Chemo-immunotherapy arm): Patients in this arm will receive standard chemotherapy in combination with a PD-1/PD-L1 inhibitor as neoadjuvant therapy prior to definitive surgery. Concomitant treatments may be administered when clinically indicated.
- ADC plus PD-1/PD-L1 inhibitor (ADC-immunotherapy arm): Patients in this arm will receive an antibody-drug conjugate (ADC) in combination with a PD-1/PD-L1 inhibitor as neoadjuvant therapy prior to definitive surgery. Concomitant treatments may be administered when clinically indicated.

SUMMARY:
This study aims to evaluate whether psychological status affects the response to neoadjuvant immunotherapy in triple-negative breast cancer (TNBC) and how it relates to immune changes during treatment. Participants will receive standard therapy, undergo psychological assessments, and provide blood and saliva samples for biomarker testing. By linking psychological status with immune profiles and treatment outcomes, the study seeks to clarify how mental state may influence immunotherapy effectiveness.

DETAILED DESCRIPTION:
The goal of this prospective observational study is to understand how psychological status influences the therapeutic response and long-term outcomes of patients with triple-negative breast cancer (TNBC) receiving neoadjuvant immunotherapy. The study primarily focuses on the association between psychological status and pathological complete response (pCR) as well as event-free survival (EFS).

In this study, early-stage TNBC patients undergoing standard neoadjuvant immunotherapy will complete psychological assessments at baseline and multiple timepoints during treatment. Measurement include self-assessment questionnaires like GAD-7 and PHQ-9 and clinician-administered depression assessment scale like Hamilton Depression Rating Scale (HDRS). Blood and saliva samples will be collected to measure immune cell subsets, inflammatory cytokines, cortisol, and heart rate variability (HRV). Treatment response (pCR, ORR) and long-term outcomes (EFS) will be recorded and analyzed. By integrating psychological measures, circulating immune markers, and clinical efficacy endpoints, researchers aim to build a psychological-immune-response association model and identify psychophysiological biomarkers that may predict immunotherapy benefit.

ELIGIBILITY:
Inclusion Criteria：

Participants must meet all of the following criteria:

1. Age ≥ 18 years;
2. Female patients;
3. Voluntarily agrees to participate in the study and signs the informed consent form, with good compliance and willingness to complete follow-up assessments;
4. Histologically confirmed invasive triple-negative breast cancer (TNBC), defined as ER < 1%, PR < 1%, and HER-2 0-1+ by IHC, or HER-2 2+ with negative FISH/CISH results (no gene amplification);
5. Planned to receive neoadjuvant immunotherapy-based treatment as part of routine clinical care.

Exclusion Criteria

Patients will be excluded if any of the following conditions apply:

1. Presence of distant metastasis;
2. History of other malignancies, except for adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or cancers with no evidence of disease for ≥ 5 years;
3. Participation in another clinical trial and receipt of an investigational drug or treatment within 30 days before initiation of neoadjuvant therapy;
4. Known immunodeficiency or HIV infection;
5. Severe cardiac, pulmonary, hepatic, or renal dysfunction;
6. Uncontrolled infection or active systemic infection;
7. Pregnancy or breastfeeding;
8. Severe psychological or cognitive impairment that precludes completion of psychological assessments.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from women diagnosed with early-stage triple-negative breast cancer who are receiving neoadjuvant immunotherapy at Fudan University Shanghai Cancer Center (FUSCC). The study population consists of both outpatient and inpatient breast cancer patients treated at this tertiary cancer referral center, which serves a large and diverse region across Shanghai and surrounding regions. Eligible participants will be enrolled prior to initiation of neoadjuvant treatment and followed throughout the perioperative period.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) Rate | At the time of definitive surgery
  Pathological complete response (pCR) is defined as the absence of residual invasive cancer in the breast and axillary lymph nodes (ypT0/Tis ypN0) after completion of neoadjuvant therapy. pCR will be assessed by investigators according to institutional pathology standards. The primary objective of this study is to evaluate the association between patients' psychological status and pCR.
Event-Free Survival (EFS) | 18 Months
  Event-free survival (EFS) is defined as the time from initiation of neoadjuvant immunotherapy until the date of one of the following events, whichever occurs first: disease recurrence, progression during neoadjuvant or adjuvant therapy, second primary malignancy, or death from any cause. Patients without an event at the end of follow-up will be censored at their last disease assessment. The study aims to investigate the relationship between baseline psychological status and long-term oncologic outcomes (EFS) in TNBC patients.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 18 Months
  Objective response rate is defined as the proportion of patients achieving a complete response (CR) or partial response (PR) to immunotherapy, as assessed by investigators according to RECIST v1.1 criteria. This outcome will be used to evaluate the association between patients' psychological status and immunotherapy response.
Correlation Between Psychological Status-Related Blood Biomarkers and Treatment Response | 18 Months
  Peripheral blood indicators that are found to be associated with psychological stress (e.g., systemic inflammation markers, cytokine signatures) will be further examined for their correlation with both pCR and ORR to explore potential psychoneuroimmune pathways mediating treatment response.
Quality of Life and Emotional Trajectory During Treatment | 18 Months
  Quality of life (QoL) and emotional changes over the course of treatment will be assessed longitudinally using validated instruments (e.g., SF-36, EORTC QLQ-C30). This outcome aims to evaluate the impact of psychological status on patients' treatment experience and well-being throughout the therapeutic course.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shangahi Cancer Center, Shanghai, Please Select, China

IPD SHARING:
Plan to Share IPD: No